CLINICAL TRIAL: NCT03200977
Title: Observational Cohort Study to Characterize the Safety of Allogeneic Hematopoietic Cell Transplantation (HCT) For Patients With Classical Hodgkin Lymphoma (CHL) Treated With Nivolumab
Brief Title: Safety of Allogeneic Hematopoietic Cell Transplantation (HCT) For Patients With Classical Hodgkin Lymphoma (CHL) Treated With Nivolumab
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-835
Record Dates: First submitted 2017-06-26; First posted 2017-06-27 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (2):
- Exposed to nivolumab prior to allogeneic HCT: patients who were treated with nivolumab-based regimen prior to an allogeneic HCT
  Interventions: Other: Non-Interventional
- Unexposed to nivolumab prior to allogeneic HCT: patients who were not treated with nivolumab-based regimen prior to an allogeneic HCT
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
An observational database analysis, using existing data of patients diagnosed with Classical Hodgkin Lymphoma.

DETAILED DESCRIPTION:
This study will include a retrospective and prospective observational database analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to18 years;
* First allogeneic HCT for cHL;
* Patients with prior autologous HCT for cHL;
* Any conditioning regimen, graft source or donor type.
* For the primary analysis additional criterion includes prior exposure to nivolumab for treatment of cHL immediately prior to the allogeneic HCT, as defined as nivolumab used alone or in combination with other agents and used as the last line of therapy prior to an allogeneic HCT with the interval between the last dose of nivolumab and start of the conditioning regimen no longer than 12 months.

Exclusion Criteria:

* Patients with nodular lymphocyte-predominant HL
* Previous chimeric antigen receptor T-cell therapy or other genetically modified cellular product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will target enrollment of 90 patients who were treated with nivolumab-based regimen prior to an allogeneic HCT with at least 45 patients who received nivolumab immediately prior to the allogeneic HCT
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Treatment-Related Mortality (TRM) | At 6 months after an allogeneic HCT
  Treatment-Related Mortality at 6 months after an allogeneic Hemaetopoietic Cell Transplantation (HCT) among patients with cHL who were previously treated with nivolumab

SECONDARY OUTCOMES:
Incidence of disease progression | Up to 2 years
  Measured by clinical assessment
Incidence of acute Graft Versus Host Disease (GVHD) | Up to 2 years
  Either Grade II-IV or Grade III-IV acute GVHD. Measured by clinical assessment
Incidence of chronic Graft Versus Host Disease (GVHD) | Up to 2 years
  Measured by clinical assessment
Incidence of post-transplant sinusoidal obstruction syndrome (SOS) | Up to 2 years
  Measured by clinical assessment
Incidence of post-transplant interstitial pneumonitis (IPN) | Up to 2 years
  Measured by clinical assessment
Incidence of post-transplant renal toxicity requiring dialysis | Up to 2 years
  Measured by clinical assessment
Overall Survival (OS) | Up to 2 years
  OS is measured from the date of allogeneic transplant to death.
Progression-Free Survival (PFS) | Up to 2 years
  PFS is measured from the date of allogeneic transplant to the date of disease progression or death.
TRM at 100 days | At 100 days after an allogeneic HCT
  Treatment-Related Mortality at 100 days after an allogeneic Hemaetopoietic Cell Transplantation (HCT) among patients with cHL who were previously treated with nivolumab
TRM at 1 year | At 1 year after an allogeneic HCT
  Treatment-Related Mortality at 1 year after an allogeneic Hemaetopoietic Cell Transplantation (HCT) among patients with cHL who were previously treated with nivolumab
TRM at 2 years | At 2 years after an allogeneic HCT
  Treatment-Related Mortality at 2 years after an allogeneic Hemaetopoietic Cell Transplantation (HCT) among patients with cHL who were previously treated with nivolumab

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Local Institution - 0001, Lawrenceville, New Jersey
  - Center for International Blood and Marrow Transplant Research, Milwaukee, Wisconsin

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html